CLINICAL TRIAL: NCT01244282
Title: A Pilot Clinical Trial to Study Arterial Spin Labeling and USPIO-enhanced MRI Methodologies for Measuring Hemodynamic Responses to Non-Drug Stimuli in Healthy Subjects
Brief Title: A Study of Two Methodologies for Measuring Blood Flow in the Brain in Response to Non-Drug Stimuli (P08085/MK-0000-180)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: P08085
Record Dates: First submitted 2010-11-17; First posted 2010-11-19 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Functional Magnetic Resonance Imaging
Keywords: brain imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Participants (Experimental): fMRI studies with sensory stimulation in the presence of 0 mg, 250 mg, 350 mg, and 510 mg cumulative doses of ferumoxytol
  Interventions: Procedure: fMRI with sensory stimulation

INTERVENTIONS:
Procedure: fMRI with sensory stimulation — BOLD fMRI study with sensory stimulation followed by fMRI in the presence of increasing concentrations of ferumoxytol (Feraheme™)

SUMMARY:
This study will identify a dose of ferumoxytol that can reliably detect changes in blood flow/volume in response to non-drug stimuli. The study will determine whether signal detection for functional magnetic resonance imaging (fMRI) using ferumoxytol is better than that for blood oxygen level-dependent (BOLD) fMRI in response to sensory stimulation. The following procedures will be conducted in each of two study periods: arterial spin labeling (ASL) imaging study with increasing exposure to carbon dioxide (CO2); BOLD fMRI study with sensory stimulation; MRI studies with sensory stimulation in the presence of increasing doses of ferumoxytol; MRI study with increasing exposure to CO2 in the presence of ferumoxytol. There will be a 3-week interval between the two study periods. The study will enroll 8 subjects, but an additional 4 subjects are permitted to enroll to preserve study power.

DETAILED DESCRIPTION:
Study Design: Translational Medicine - Imaging Platform Development

ELIGIBILITY:
Inclusion Criteria:

* Participant weighs approximately 55-75 kg and has a Body Mass Index (BMI) of 18-25 kg/m^2
* Participant is in good health
* Participant is a nonsmoker and/or has not used nicotine or nicotine-containing products for at least 6 months

Exclusion Criteria:

* Participant has a contraindication to MRI including cardiac pacemaker, brain aneurysm clip, implanted neurostimulator, insulin pump, cochlear implant, metal slivers in the eyes, or any other MRI-incompatible metal implants that cannot be safely removed
* Participant has a condition that would limit his ability to complete MRI procedures, such as claustrophobia or chronic back pain
* Participant plans to undergo MRI studies in the 3 months following the post-study visit
* Participant has a history of hemochromatosis or other conditions of iron overload or disease of iron metabolism
* Participant has a known sensitivity to ferumoxytol or iron-containing products or has a history of severe allergies, anaphylactic reaction, or intolerance to drugs and/or foods
* Participant has a history of stroke, chronic seizures, or major neurological disorder
* Participant is unable to refrain from the use of any medication, including prescription and non-prescription drugs or herbal remedies from approximately 2 weeks prior to the first dose of ferumoxytol until the post-study visit
* Participant has a history of significant head injury/trauma with loss of consciousness lasting for 15 minutes and one or more of the following: a) recurring seizures resulting from head injury; b) persistent neurological or cognitive sequelae of the injury; c) cognitive rehabilitation following the injury

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-11; Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Magnitude of the MRI percent signal change in response to sensory stimulation without administration of ferumoxytol (BOLD fMRI) | 45 minutes after initiation of imaging procedures
Magnitude of the MRI percent signal change in response to sensory stimulation following administration of the first dose of ferumoxytol (250 mg) | 55 minutes after initiation of imaging procedures
Magnitude of the MRI percent signal change in response to sensory stimulation following administration of the second dose of ferumoxytol (100 mg, total cumulative dose of 350 mg) | 70 minutes after initiation of imaging procedures
Magnitude of the MRI percent signal change in response to sensory stimulation following administration of the third dose of ferumoxytol (180 mg, total cumulative dose of 510 mg) | 85 minutes after initiation of imaging procedures